CLINICAL TRIAL: NCT01918774
Title: Cognitive Behavioral Therapy to Enhance Competitive Work Outcomes
Brief Title: Cognitive Behavior Therapy for Work Success in Veterans With Mental Illness: A Pre-post Efficacy Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: D0943-W
Record Dates: First submitted 2013-08-05; First posted 2013-08-08 (Estimated); Results first posted 2019-08-19 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-07

CONDITIONS: Mental Disorders; Mental Health Services
Keywords: Unemployment; Cognitive Behavioral Therapy; Mental Disorders
MeSH Terms: conditions — Mental Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cognitive behavior therapy for work success (Other): Fifty participants will take part in the 12 week CBTw program. All participants will receive standard SE services during the study. The longitudinal design will consist of assessments of competitive employment outcomes, important psychosocial outcomes, and background and demographic variables at baseline and at two follow-up periods' immediately following the conclusion of the CBTw program and six months after the conclusion of the program.
  Interventions: Behavioral: Cognitive behavior therapy for work success (CBTw)

INTERVENTIONS:
Behavioral: Cognitive behavior therapy for work success (CBTw) — The CBTw program includes 12 sessions that are delivered in a weekly one-hour group format. Sessions focused on identifying and modifying maladaptive thoughts related to work, enhancing self efficacy and beliefs in one's ability to succeed at work, identifying and addressing personal barriers to work, and increasing beneficial coping strategies that can be applied across employment settings, including during the job search phase and working on the job. The intervention is tailored toward both employed and unemployed persons seeking community work. Session content includes the following modules: Introduction-Work goals and work story; CBT model and work; Thinking about work; Barriers to work; Coping with stress and anxiety; Coping with anger and difficult emotions; Communication at work; Dealing effectively with people at work; Managing work success; Personal work success plan.

SUMMARY:
In 2010, 11.5% of all Gulf War-II Veterans were unemployed; that figure rose to 15.2% in January 2011 and continues to grow as the number of Veterans from recent wars increases. The prevalence of mental illness among Veterans is also notable; estimates range from 31% to nearly 37% for any psychiatric disorder, and over half of these Veterans are diagnosed with more than one psychiatric condition. In addition, empirical evidence suggests that some mental disorders are more prevalent in Veterans than in the general population. Linking unemployment and mental illness, a recent study found that 65% of Veterans using VA healthcare were unemployed, and compared to employed Veterans, the unemployed were more likely to have depression, bipolar disorder, post traumatic stress disorder (PTSD), schizophrenia, or substance use disorders. Vocational dysfunction was reported most often in disabled Veterans with schizophrenia, PTSD, and substance use disorders. Not surprisingly, this study also found that unemployed Veterans had significantly lower income than employed persons. Similarly, a large study focusing specifically on Veterans with PTSD concluded that vocational dysfunction is a notable problem among this group, as they were significantly less likely to be employed after participating in VA work programs compared with participants without the disorder. Because most individuals with mental illness desire to work in regular competitive employment, the nationwide problem of unemployment among Veterans with mental illness is particularly troubling.

The VA is addressing this need by implementing supported employment (SE), a psychiatric rehabilitation approach that provides individual vocational assistance to Veterans with mental illness. While the SE model is empirically validated and SE programs have been shown to achieve partial success in improving employment outcomes, a sizable proportion of individuals, 40% or more, remain unemployed. A further challenge is job retention; Veterans with mental illness who obtain jobs frequently struggle to maintain them long-term. Even in the context of high quality, evidence-based vocational services, most studies show only modest job retention of a few months, and consequently, frequent job losses and inconsistent vocational functioning remain a substantial and unsolved problem.

Rationale: Cognitive behavioral therapy (CBT) effectively reduces symptoms across a range of psychiatric conditions; however, its benefit to functioning remains less well understood. Work functioning has received little empirical attention in the CBT domain. Despite research evidence suggesting that maladaptive thoughts about oneself and expectations about the ability to work interfere with work success, no CBT programs have been developed specifically targeting vocational themes with the goal of improving competitive work outcomes. Further, a recent paper outlined needed avenues of future study in the SE domain; Drake and Bond (2011) state that cognitive strategies may be a fruitful area to develop to help "nonresponder" consumers with mental illness who struggle with vocational dysfunction despite high quality vocational assistance. The goal of the current project is to address this gap and the serious problem of unemployment in Veterans with mental illness by pilot testing the CBT for work success program (CBTw) and assessing key employment outcomes before and after the intervention, and six months after conclusion of the intervention.

Specific Aims:

Aim 1: Test the preliminary efficacy of the CBTw program on key Veteran employment and psychosocial outcomes utilizing a pre/post design.

Aim 2: Further assess the feasibility of the program, including recruitment, retention rates, and program participation rates.

Aim 3: Gauge effect sizes in preparation for a larger randomized controlled trial examining the effectiveness of the CBT program in routine practice settings

DETAILED DESCRIPTION:
Background and Significance In 2010, 11.5% of all Gulf War-II Veterans were unemployed; that figure rose to 15.2% in January 2011 and continues to grow as the number of Veterans from recent wars increases. The prevalence of mental illness among Veterans is also notable; estimates range from 31% to nearly 37% for any psychiatric disorder, and over half of these Veterans are diagnosed with more than one psychiatric condition. In addition, empirical evidence suggests that some mental disorders are more prevalent in Veterans than in the general population. Linking unemployment and mental illness, a recent study found that 65% of Veterans using VA healthcare were unemployed, and compared to employed Veterans, the unemployed were more likely to have depression, bipolar disorder, post traumatic stress disorder (PTSD), schizophrenia, or substance use disorders. Vocational dysfunction was reported most often in disabled Veterans with schizophrenia, PTSD, and substance use disorders. Not surprisingly, this study also found that unemployed Veterans had significantly lower income than employed persons. Similarly, a large study focusing specifically on Veterans with PTSD concluded that vocational dysfunction is a notable problem among this group, as they were significantly less likely to be employed after participating in VA work programs compared with participants without the disorder. Because most individuals with mental illness desire to work in regular competitive employment, the nationwide problem of unemployment among Veterans with mental illness is particularly troubling.

The VA is addressing this need by implementing supported employment (SE), a psychiatric rehabilitation approach that provides individual vocational assistance to Veterans with mental illness. While the SE model is empirically validated and SE programs have been shown to achieve partial success in improving employment outcomes, a sizable proportion of individuals, 40% or more, remain unemployed. A further challenge is job retention; Veterans with mental illness who obtain jobs frequently struggle to maintain them long-term. Even in the context of high quality, evidence-based vocational services, most studies show only modest job retention of a few months, and consequently, frequent job losses and inconsistent vocational functioning remain a substantial and unsolved problem. In response to this problem, it has been suggested that interventions focusing on patient-level barriers augment existing vocational services.

Rationale Cognitive behavioral therapy (CBT) effectively reduces symptoms across a range of psychiatric conditions; however, its benefit to functioning remains less well understood. Some studies have evidenced a positive influence of CBT on functional outcomes, whereas others have not. One possible explanation for these inconsistencies across studies is that CBT interventions are most often focused on symptoms rather than community functioning. The few CBT interventions that have been specifically designed to address functioning have shown promising results. One functional area of critical importance is work-a central goal of most Veterans with (and without) mental illness. However, work functioning has received little empirical attention in the CBT domain. Despite research evidence suggesting that maladaptive thoughts about oneself and expectations about the ability to work interfere with work success, no CBT programs have been developed specifically targeting vocational themes with the goal of improving competitive work outcomes. Further, a recent paper outlined needed avenues of future study in the supported employment domain; Drake and Bond (2011) state that cognitive strategies may be a fruitful area to develop to help "nonresponder" consumers with mental illness who struggle with vocational dysfunction despite high quality vocational assistance. The goal of the current project is to address this gap and the serious problem of unemployment in Veterans with mental illness by testing a CBT program designed to enhance competitive work functioning in this population.

Aim 1: Test the preliminary efficacy of the CBTw program on key Veteran employment and psychosocial outcomes utilizing a pre/post design.

Aim 2: Further assess the feasibility of the program, including recruitment, retention rates, and program participation rates.

Aim 3: Gauge effect sizes in preparation for a larger randomized controlled trial examining the effectiveness of the CBT program in routine practice settings

Research Design and Methods This study will pilot test a cognitive behavior therapy (CBT) intervention for persons with mental illness to target improved competitive employment outcomes, termed the "CBT for Work Success (CBTw) program"; this CBT intervention will serve as a compliment to existing supported employment services in the VA. Fifty participants will take part in the 12 week group-based CBTw program. All participants will receive standard SE services during the study. The longitudinal design will consist of assessments of competitive employment outcomes, important psychosocial outcomes, and background and demographic variables at baseline and at two follow-up periods-immediately following the conclusion of the CBTw program and six months after the conclusion of the program.

Measures Unless otherwise specified, study measures will be collected at three time points: baseline, post intervention, 3 month follow up.

Background Characteristics. Collected at baseline only, participant background characteristics will include sex, age, ethnicity, educational attainment, mental health diagnosis, marital status, residential status, current work status (employed/unemployed), work history (i.e., weeks worked during the six months preceding the study; legal history. The investigators will collect this data through a combination of SE records, patient medical records (i.e., CPRS), and participant self-report.

Competitive Employment Outcomes. Competitive employment outcomes will be assessed at the two follow-up time points (after the intervention and 6 month follow-up) through participant self-report and supported employment records when available. These outcomes are standard in studies of employment in persons with mental illness and will include employment status (working/not working), job acquisition rate, total number of job losses, the total and mean number of weeks worked over the follow-up period, job tenure defined as achievement of steady competitive work--working at least half the follow up period (6 month follow up only), and total and mean wages earned across the study and follow-up periods.

Work-related self-efficacy. Work related self-efficacy is defined as one's perceived ability and confidence to perform work activities. Given that the adapted CBT program will seek to improve these perceptions, the investigators will measure this construct using the Work-Related Self-efficacy Scale. The 37-item self-report scale yields a total score and measures four sub-domains of self-efficacy: general work skills, career planning, job securing skills, and work-related social skills. Studies suggest that the scale has adequate to good reliability and validity in adults with mental illness living in the community.

Motivation to work: Motivation to work will be measured by the Work Extrinsic and Intrinsic Motivation Scale (WEIMS) based on self determination theory; the 18-item WEIMS measures six empirically grounded domains of motivation, including 1). intrinsic motivation (e.g., "I want to work for the satisfaction I experience from taking on interesting challenges"); 2). integrated regulation motivation (e.g., I want to work because it is a fundamental part of who I am."); 3) identified regulation motivation (e.g., "I want to work to attain a certain lifestyle"; 4) introjected regulation (e.g., "I want to work because I want to be a winner in life."); 5) external regulation (e.g., I want to work because it provides me with security."); 6) amotivation (e.g., "I don't know why I want to work."). The WEIMS is scored on a 1 to 7 Likert scale ('Does not correspond at all' to 'Corresponds exactly') with higher scores indicating higher levels of each domain of motivation. The WEIMS has been shown to have strong predictive validity, correlating highly with work behaviors.

Global motivation to work will be measured with one item: "How motivated are you to work?" measured on a 1 to 10 Likert scale, 1-'Not at all motivated'; 10-'Extremely motivated'.

Work effectiveness & Work Productivity. The Work and Health Interview will assess work effectiveness and work productivity for participants who are currently working (unemployed participants will not complete these measures). Work effectiveness will be measured by one self-report item-" On days that you worked during the past 4 weeks, how effective were you in your job on average? Please tell me, on a scale of 0 to 100, where 0% means that you were not at all effective, and 100% means that you were completely effective, how effective would you say you have been on your job during the past 4 weeks?" Work productivity will be measured by 7 self-report items scored on a Likert scale ranging from 0, "none of the time" to 4, "all the time" (item example: "Work more slowly than usual?"). Participants will report on work productivity over the last two weeks. The Work and Health Interview has been used widely in patients with chronic conditions, demonstrating good psychometric properties.

Self-esteem: The Rosenberg self esteem scale (RSES), a 10-item Likert scale (1-strongly agree; 2-agree; 3-disagree; 4-strongly disagree) will examine self esteem; higher scores on the RSES indicate higher levels of a unidimensional self-esteem construct. The RSES has been used extensively in samples of persons with and without mental illness and across various ethnic and cultural groups, demonstrating good reliability and validity.

Quality of Life. Prior studies in the mental health domain have demonstrated that quality of life improves in response to CBT treatment, therefore, as discussed above with regard to symptoms, quality of life may be enhanced in response to CBT treatment, regardless of the impact on work outcomes. The Quality of Life Interview (QOLI), developed specifically for a psychiatric population, will measure Veteran quality of life. The investigators will use the 17 items that assess subjective quality of life, including global life satisfaction and the following sub-domains: living situation, daily activities and functioning, family relations, social relations, legal and safety issues, and health. The QOLI has been shown to have very good reliability and validity in adult outpatients.

Subjective Recovery: Global perceived recovery will be assessed by the Recovery Assessment Scale (RAS), a 41 item scale designed to assess perceptions of recovery held by persons with mental illness. Because perceptions of recovery may be amenable to CBT and have been associated with key functional outcomes, including employment, it is appropriate to examine in this study. The self-report RAS is scored on a 1 to 5 Likert scale from 'strongly disagree' to 'strongly agree' (e.g., "I have a desire to succeed."). The RAS has five factors including "confidence and hope," "willingness to ask for help", "goal and success orientation", "reliance on others", and "no domination by symptoms." Higher scores indicate stronger held perceptions of personal recovery. The RAS has shown good test retest reliability, internal consistency, and criterion-related validity.

Symptoms. Symptoms are essential to assess in this study, as they are often the primary beneficiary of CBT intervention, demonstrating moderate to large effect sizes in randomized trials across numerous psychiatric conditions. Thus, it is possible that symptoms may improve in response to CBT treatment, regardless of change in employment status.

Psychiatric symptoms often present in schizophrenia-spectrum disorders will be assessed by the Positive and Negative Syndrome Scale (PANSS), which has been used extensively in studies of psychiatric rehabilitation and CBT. The PANSS is comprised of 30 items scored on a 1 to 7 Likert scale, in which the total score is obtained by adding up scores on all 30 items (total scores range from 30 to 240). The PANSS has five subscales identified via factor analytic studies including the Positive syndrome (6 items), Negative syndrome (8 items), Emotional discomfort (4 items), Hostility (4 items), and Cognitive (7 items). The PANSS has adequate reliability and validity.

In addition, the investigators will assess depression and anxiety, two commonly occurring psychiatric conditions in Veterans; depression and anxiety are linked with vocational dysfunction and have been demonstrated to respond well to CBT. Current levels of depression will be assessed using the Beck Depression Inventory, Second Edition. The BDI-II contains 21 items that assess the various mood and bodily symptoms of depression; participants are asked to respond based on symptoms during the past two weeks. There are four response options for each item reflecting increasing severity of depression; the total score is obtained by summing up the scores on each item (0-3). The BDI-II is the gold standard tool to assess depression in both non-clinical and psychiatric populations and has been shown to have excellent reliability and validity across several prior studies.

Thirdly, symptoms of anxiety will be assessed using the Beck Anxiety Inventory. The BAI has 21 items, each describing a psychological or physiological symptom of anxiety (e.g., "Nervous") that respondents rate on a 0 to 3 Likert Scale ("not at all" to "severely") based on how much they have been bothered by the symptom within the past week. The BAI has been widely used to assess anxiety in adults with mental illness and has been demonstrated to have strong psychometric properties.

Current substance use will be assessed at baseline; this in consideration of the investigators' previous work demonstrating a link between active substance use and difficulties obtaining work for Veteran with mental illness receiving SE services. In addition, substance abuse may hinder participants from benefiting from the CBTw intervention. The investigators will use the recent substance use section of the Addiction Severity Index (ASI), which assesses use of a variety of substances in the previous 30 days.

Feasibility Assessment: Feasibility of the CBTw program will be assessed by evaluating the following recruitment, retention, and participation outcomes during the CBTw pilot and at the follow-up periods: (1) number of participants who are enrolled in the study, (2) number who attend 50% or more of group sessions, indicating adequate "exposure" to the program, (4) mean number of sessions attended; (5) number of participants who complete post-treatment follow-up assessments, and (6) number of participants who complete 6-month follow-up assessments; 7) number of participants who dropout of the CBTw program.

Fidelity to cognitive behavioral therapy: Adherence to the CBT model will be assessed by an adapted form of the Revised Cognitive Therapy Scale (CTS-R). The group therapy version is comprised of seven items rated on a 0-6 likert scale, with rating of "3" or greater on each item indicating fully-competent practice compared to the average skilled clinician. Prior studies using the group therapy version of the CTS-R has found good to excellent interrater reliability. Furthermore, fidelity will be assessed using audio recordings of three random sessions per CBTw group and will be conducted by a blinded member of the study team trained in CBT fidelity by Dr. Kukla.

Analysis Data will be analyzed using the Statistical Package for the Social Sciences (SPSS), version 20. First, frequency distributions and histograms will be generated to determine the normality of the sampling distribution and inspect for outliers. If the distribution is skewed, data transformations and the use of nonparametric tests in primary analyses will be considered. Secondly, descriptive statistics will be generated to characterize the demographic and background composition of the sample and levels of outcome variables at baseline, post-treatment, and three months post-treatment. This mean and standard deviation information obtained will be used for sample size calculation for a future expanded randomized trial.

Next, study outcomes will be compared between baseline and the two follow up time points using a series of dependent groups T-tests. Significance values for t-tests will be set at p<.025 to account for the effect of inflated alpha due to multiple comparisons. Next, mixed effects regression models will be conducted including a random effect to account for the nested nature of the data, (i.e. three measurement points nested within participant). These models will identify of trajectories of change in outcomes over time and will allow for the inclusion of important covariates (e.g., employment history assessed at baseline). P values will be set at .05.

Clinical Significance Information from this study will help guide the activities in future planned studies. Specifically, this will lead to a future larger VA merit study testing the intervention using a randomized controlled design that is scalable to routine service settings.

ELIGIBILITY:
Inclusion Criteria:

* Participants include Veterans who are receiving individualized vocational services at an urban Midwestern VA medical center.
* Inclusion criteria are a diagnosis of a mental disorder as confirmed through medical record review, current enrollment in vocational services, and an active goal of working in the community

  * participants may be currently working in the community or unemployed and searching for work

Exclusion Criteria:

* Exclusion criteria is a major cognitive deficit or severe medical condition that would prevent participation in the intervention and/or competitive community work.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marina Elizabeth Kukla, BS MS PhD, Principal Investigator — Richard L. Roudebush VA Medical Center, Indianapolis, IN
Locations (1):
- Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kukla M, McGuire AB, Salyers MP. Rural and urban supported employment programs in the Veterans Health Administration: Comparison of barriers and facilitators to vocational achievement for veterans experiencing mental illnesses. Psychiatr Rehabil J. 2016 Jun;39(2):129-36. doi: 10.1037/prj0000184. Epub 2016 Apr 7. PMID 27054902
- [Result] Kukla M, McGuire AB, Salyers MP. Barriers and Facilitators Related to Work Success for Veterans in Supported Employment: A Nationwide Provider Survey. Psychiatr Serv. 2016 Apr 1;67(4):412-7. doi: 10.1176/appi.ps.201500108. Epub 2015 Dec 15. PMID 26695496
- [Result] Kukla M, Strasburger AM, Lysaker PH. A CBT Intervention Targeting Competitive Work Outcomes for Persons With Mental Illness. Psychiatr Serv. 2016 Jun 1;67(6):697. doi: 10.1176/appi.ps.670504. No abstract available. PMID 27245085
- [Result] Kukla M, Strasburger AM, Salyers MP, Rattray NA, Lysaker PH. Subjective Experiences of the Benefits and Key Elements of a Cognitive Behavioral Intervention Focused on Community Work Outcomes in Persons With Mental Illness. J Nerv Ment Dis. 2017 Jan;205(1):66-73. doi: 10.1097/NMD.0000000000000601. PMID 27741081
- [Result] Kukla M, Strasburger AM, Salyers MP, Rollins AL, Lysaker PH. A Pilot Test of Group Based Cognitive Behavioral Therapy to Augment Vocational Services for Persons With Serious Mental Illness: Feasibility and Competitive Work Outcomes. J Nerv Ment Dis. 2018 May;206(5):310-315. doi: 10.1097/NMD.0000000000000796. PMID 29485477
- [Result] Kukla M, Salyers MP, Strasburger AM, Johnson-Kwochka A, Amador E, Lysaker PH. Work-focused cognitive behavioral therapy to complement vocational services for people with mental illness: Pilot study outcomes across a 6-month posttreatment follow-up. Psychiatr Rehabil J. 2019 Dec;42(4):366-371. doi: 10.1037/prj0000365. Epub 2019 May 9. PMID 31070442

RESULTS

PARTICIPANT FLOW:
Groups:
- Cognitive Behavioral Therapy for Work Success: Adults with mental illness who are receiving vocational services and have a competitive work goal will take part in the 12-session Cognitive Behavioral Therapy for Work Success (CBTw) intervention. CBTw is a group-based intervention that occurs weekly (1 hour group sessions) for 12 weeks.
Period: Overall Study
Arm/Group | Cognitive Behavioral Therapy for Work Success
Started | 57
Completed | 52
Not Completed | 5
Not completed — Lost prior to first CBTw session | 4
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Study completers
Arm/Group | Cognitive Behavioral Therapy for Work Success
Number analyzed (Participants) | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 30
  African American/Black | 22
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 52
Mental Health Diagnosis [Count of Participants; unit: Participants]
  Schizophrenia Spectrum Disorders | 20
  Mood disorders | 21
  Anxiety disorders | 7
  Posttraumatic stress disorder | 4
Educational Attainment [Count of Participants; unit: Participants]
  High school/GED | 13
  Some college or technical school (no degree) | 26
  Associate's degree | 1
  Bachelor's degree | 9
  Master's degree | 3
Current work status [Count of Participants; unit: Participants]
  Unemployed at baseline | 44
  Employed at baseline | 8
Marital status [Count of Participants; unit: Participants]
  Married | 6
  Unmarried | 46
Residential Status [Count of Participants; unit: Participants]
  Independent living | 28
  Supportive housing | 13
  Non-independent living | 11
Work history-weeks employed in 6 months preceding baseline [Mean (Standard Deviation); unit: weeks] | 3.9 (8.0)
Legal history-felony convictions [Count of Participants; unit: Participants]
  felony convictions | 16
  no felony convictions | 36

OUTCOME MEASURES:

1. Primary Outcome: Change in Competitive Employment
Description: Competitive employment is standard in studies of employment in persons with mental illness and will include change in the total number of weeks worked in competitive jobs between baseline and the 6 month follow-up point.
Time Frame: Change from baseline competitive employment to 6 month follow up competitive employment
Population: Open trial treatment, all participants who completed the study are included.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Cognitive Behavioral Therapy for Work Success
Number analyzed (Participants) | 52
weeks | 13.6 (11.2)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy for Work Success; Test type: Other — Pre-post analysis comparing weeks worked in the 6 months preceding baseline and the 6 month study follow-up; p < .001, within groups t-test — A priori threshold of significance was p<.05

2. Primary Outcome: Number of Participants With Steady Competitive Work Attainment
Description: Steady competitive work attainment, defined as working at least half the follow up period, will be assessed at the 6 month follow up.
Time Frame: 6 month follow up
Population: All participants who completed the study are included in analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Cognitive Behavioral Therapy for Work Success
Number analyzed (Participants) | 52
Participants | 27

3. Secondary Outcome: Work Effectiveness
Description: The Work and Health Interview (Stewart et al., 2003) will assess work effectiveness and work productivity for participants who are currently working (unemployed participants will not complete these measures). Work effectiveness will be measured by one self-report item-" On days that you worked during the past 4 weeks, how effective were you in your job on average? Please tell me, on a scale of 0 to 100, where 0% means that you were not at all effective, and 100% means that you were completely effective, how effective would you say you have been on your job during the past 4 weeks?". Higher scores indicate more work effectiveness. The Work and Health Interview has been used widely in patients with chronic conditions, demonstrating good psychometric properties.
Time Frame: baseline and 12 week follow up scores
Population: Participants who worked in competitive jobs during the 12 week follow up were included.
Measure: Mean (Standard Deviation); unit: percentage of work effectiveness score
Arm/Group | Cognitive Behavioral Therapy for Work Success
Number analyzed (Participants) | 30
percentage of work effectiveness score
  baseline score | 46.9 (47.3)
  12 week follow up score | 88.7 (13.2)

4. Secondary Outcome: Positive and Negative Syndrome Scale (PANSS)
Description: The Positive and Negative Syndrome Scale (PANSS) has been used extensively in studies of psychiatric rehabilitation and CBT. The PANSS (Kay et al., 1987) is comprised of 30 items scored on a 1 to 7 Likert scale, in which the total score is obtained by adding up scores on all 30 items (total scores range from 30 to 240). Higher scores indicate more severe symptoms. The PANSS has adequate reliability and validity in adults with severe mental illness (Kay et al., 1987).
Time Frame: baseline, 12 week follow up
Population: Participants who completed the study were included.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Behavioral Therapy for Work Success
Number analyzed (Participants) | 52
score on a scale
  baseline score | 57.9 (11.2)
  12 week follow up score | 57.3 (15.3)

5. Secondary Outcome: Beck Depression Inventory (BDI-II)
Description: Change in levels of depression will be assessed using the Beck Depression Inventory, Second Edition (BDI-II; Beck, Steer, & Brown, 1996). The BDI-II contains 21 items that assess the various mood and bodily symptoms of depression; participants are asked to respond based on symptoms during the past two weeks. There are four response options for each item reflecting increasing severity of depression; the total score is obtained by summing up the scores on each item (0-3). Total scores range from 0 to 63, with higher scores indicating more severe depressive symptoms. The BDI-II is the gold standard tool to assess depression in both non-clinical and psychiatric populations and has been shown to have excellent reliability and validity across several prior studies (e.g., Yin & Fan, 2000).
Time Frame: baseline, post intervention (12 weeks)
Population: All participants who completed the intervention are included in the analysis
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Cognitive Behavioral Therapy for Work Success
Number analyzed (Participants) | 52
score on scale
  baseline score | 16.6 (10.3)
  12 week follow up score | 12.5 (9.7)

6. Secondary Outcome: Beck Anxiety Inventory (BAI)
Description: Symptoms of anxiety will be assessed using the Beck Anxiety Inventory (Beck & Steer, 1993). The BAI has 21 items, each describing a psychological or physiological symptom of anxiety (e.g., "Nervous") that respondents rate on a 0 to 3 Likert Scale ("not at all" to "severely") based on how much they have been bothered by the symptom within the past week. Total scores range from 0 to 63 with higher scores indicating more severe anxiety symptoms. The BAI has been widely used to assess anxiety in adults with mental illness and has been demonstrated to have strong psychometric properties (e.g., Fydrich, Dowdall, & Chambless, 1992).
Time Frame: baseline, 12 week follow up
Population: Participants who completed the study were included.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Behavioral Therapy for Work Success
Number analyzed (Participants) | 52
score on a scale
  baseline | 14.1 (10.3)
  12 week follow up | 12.6 (11.8)

7. Secondary Outcome: Work Related Self-efficacy Scale
Description: Work related self-efficacy is defined as one's perceived ability and confidence to perform work activities. Given that the adapted CBT program will seek to improve these perceptions, the investigators will measure this construct using the Work-Related Self-efficacy Scale (Waghorn et al., 2005). The 37-item self-report scale yields a total score on a 0 to 100 point scale, in which higher scores indicate stronger self efficacy related to work. Studies suggest that the scale has adequate to good reliability and validity in adults with mental illness living in the community (Harris et al., 2010).
Time Frame: baseline, 12 week follow up
Population: Participants who completed the study are included.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Behavioral Therapy for Work Success
Number analyzed (Participants) | 52
score on a scale
  baseline score | 78.7 (13.6)
  12 week follow up score | 81.0 (13.3)

8. Secondary Outcome: Quality of Life Interview
Description: Prior studies in the mental health domain have demonstrated that quality of life improves in response to CBT treatment, therefore, as discussed above with regard to symptoms, quality of life may be enhanced in response to CBT treatment, regardless of the impact on work outcomes. The Quality of Life Interview (QOLI; Lehman, 1988), developed specifically for a psychiatric population, will measure veteran quality of life. The investigators will use the 17 items that assess subjective quality of life, including global life satisfaction and sub-domains--living situation, daily activities and functioning, family relations, social relations, legal and safety issues, and health. The QOLI has been shown to have very good reliability and validity in adult outpatients (Lehman, 1988; Lehman et al., 1993). This study focused on the health quality of life domain, comprised of 6 items scores on a 1 to 7 likert scale. Scores range from 6 to 42 with higher scores indicating higher quality of life.
Time Frame: baseline, 12 week follow up
Population: Participants who completed the study were included.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Behavioral Therapy for Work Success
Number analyzed (Participants) | 52
score on a scale
  baseline score | 24.0 (4.1)
  12 week follow up score | 25.8 (5.1)

9. Secondary Outcome: Work Extrinsic and Intrinsic Motivation Scale
Description: Motivation to work will be measured by the Work Extrinsic and Intrinsic Motivation Scale (WEIMS) based on self determination theory; the 18-item WEIMS measures six empirically grounded domains of motivation, including 1). intrinsic motivation; 2). integrated regulation motivation; 3) identified regulation motivation; 4) introjected regulation; 5) external regulation ; 6) amotivation . The WEIMS is scored on a 1 to 7 Likert scale ('Does not correspond at all' to 'Corresponds exactly'). Mean WEIMS scores range from 1 to 7 with higher scores indicating higher levels of motivation. The WEIMS has been shown to have strong predictive validity, correlating highly with work behaviors (e.g., Tremblay et al., 2009).
Time Frame: baseline, 12 week follow up
Population: Participants who completed the study were included.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Behavioral Therapy for Work Success
Number analyzed (Participants) | 52
score on a scale
  baseline score | 5.7 (0.7)
  12 week follow up score | 5.6 (0.8)

10. Secondary Outcome: Rosenberg Self Esteem Scale
Description: The Rosenberg self esteem scale, a 10-item Likert scale (1-strongly agree; 2-agree; 3-disagree; 4-strongly disagree) will examine self esteem (Rosenberg, 1965); higher scores on the RSES indicate higher levels of a unidimensional self-esteem construct. The RSES has been used extensively in samples of persons with and without mental illness and across various ethnic and cultural groups, demonstrating good reliability and validity (e.g. Link et al., 2014). Scores range from 10 to 40, with lower scores indicate higher self esteem.
Time Frame: baseline to 12 week follow up
Population: All participants who completed the study are included.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Behavioral Therapy for Work Success
Number analyzed (Participants) | 52
score on a scale
  baseline score | 21.7 (4.7)
  12 week follow up score | 20.1 (5.0)

11. Secondary Outcome: Recovery Assessment Scale
Description: Global perceived recovery will be assessed by the Recovery Assessment Scale (Corrigan et al., 1999), a 41 item scale designed to assess perceptions of recovery held by persons with mental illness. Because perceptions of recovery may be amenable to CBT and have been associated with key functional outcomes, including employment, it is appropriate to examine in this study. The self-report RAS is scored on a 1 to 5 Likert scale from 'strongly disagree' to 'strongly agree' (e.g., "I have a desire to succeed."). The RAS has five factors including "confidence and hope," "willingness to ask for help", "goal and success orientation", "reliance on others", and "no domination by symptoms." Total scores range from 41 to 205, with higher scores indicating stronger perceptions of personal recovery. The RAS has shown good test retest reliability, internal consistency, and criterion-related validity (Corrigan et al., 1999).
Time Frame: baseline to 12 week follow up
Population: All participants who completed the study are included.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Behavioral Therapy for Work Success
Number analyzed (Participants) | 52
score on a scale
  baseline scores | 128.4 (12.0)
  12 week follow up scores | 133.3 (15.0)

12. Secondary Outcome: Work Productivity
Description: The Work and Health Interview (Stewart et al., 2003) will assess work productivity for participants who are currently working. Work productivity will be measured by 7 self-report items (e.g., "During the past 2 weeks, how often did you lose concentration at work?") scored on a Likert scale ranging from 0, "none of the time" to 4, "all the time" . Total scores are calculated using the mean of all items and then converted to quarter percentages, yielding a final work productivity score ranging from 0 to 100. Higher scores indicate more disruption and lower work productivity. Lower scores indicate less work disruption and higher work productivity. The Work and Health Interview has been used widely in patients with chronic conditions, demonstrating good psychometric properties.
Time Frame: baseline to 12 week follow-up
Population: Those who obtained competitive work during the 12 week follow up period
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Cognitive Behavioral Therapy for Work Success
Number analyzed (Participants) | 22
score on scale
  baseline score | 19.6 (12.1)
  12 week follow up score | 12.2 (9.7)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the 12 weeks of active study participation.
Arm/Group | Cognitive Behavioral Therapy for Work Success
All-Cause Mortality (participants affected / at risk) | 0/52
Serious Adverse Events (participants affected / at risk) | 0/52
Other Adverse Events (participants affected / at risk) | 0/52

LIMITATIONS AND CAVEATS:
Limitations of the study include a small sample size and an open trial design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-26): https://cdn.clinicaltrials.gov/large-docs/74/NCT01918774/Prot_SAP_000.pdf